CLINICAL TRIAL: NCT00507247
Title: Phase II, Open-Label Study to Evaluate the Safety and Efficacy of Daptomycin in the Treatment of Catheter-Related Staphylococcus Aureus Bloodstream Infections
Brief Title: Daptomycin in the Treatment of Catheter-Related Staphylococcus Aureus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0622; NCI-2010-00722 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2014-11

CONDITIONS: Staphylococcus Aureus
Keywords: Catheter-Related Infection; Bloodstream Infections; Staphylococcus Aureus; Daptomycin
MeSH Terms: conditions — Staphylococcal Infections; Catheter-Related Infections; Sepsis | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daptomycin (Experimental): 6mg/kg/day intravenous (IV) for 10 days
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — 6mg/kg/day IV for at least 10 days.
  Other Names: Cubicin

SUMMARY:
Primary Objective:

Evaluate the efficacy and safety of daptomycin given for treatment of catheter-related bloodstream infections due to S. aureus bacteria with or without exchange of the central venous catheter (CVC) over guide wire in comparison with a historical control group of catheter-related S. aureus bacteremia treated with standard therapy (Vancomycin) or other active agents against staph aureus (such as beta-lactam antibiotics).

DETAILED DESCRIPTION:
Daptomycin is a new antibiotic. It may be effective against a variety of bacterial infections that are difficult to treat.

Aztreonam, Cefepime, Carbapenems and Augmentin are antibiotics that are used to treat certain types of bacteria.

If you are found to be eligible to take part in this study, you will be given daptomycin by vein for at least 10 days, depending on your certain type of bacteria. You will receive Daptomycin by vein for 30 minutes every 24 hours.

The CVC associated with CRBSI (catheter-related bloodstream infection = CR-BSI) from all enrolled patients will either be removed or be exchanged over guide wire for a new CVC within 96 hours of onset of the first blood culture. Your primary doctor will decide whether to remove or exchange the CVC with the willingness of you.

If the study doctor and/or your primary physician knows or thinks that you have a mixed infection (both "gram positive" and "gram negative") or may have infection in lungs (pneumonia), you may also be treated with the antibiotic drugs Aztreonam, Cefepime, Carbapenems, or Augmentin by vein or by mouth in combination with the study drug Daptomycin.

During each week of treatment, blood (about 1 tablespoon) will be drawn for routine lab tests. The blood sample may be drawn from the CVC, if the CVC is still in place. In addition, blood (about 1 tablespoon) will be drawn every other day until it no longer shows signs of infection. The catheter exit site may be examined at each visit until you have no more signs or symptoms of infection. If you are discharged from the hospital before completing the study medication, arrangements will be made to provide infusions on an out-patient basis or home infusion.

During each week of treatment, you will be asked about any symptoms or illnesses that you have experienced. In addition, you will be asked to inform the study doctor and/or study staff of any medications or therapies that you are taking while on study. You will be taken off study if the infection gets worse or intolerable side effects occur.

Participation on this study will last for a no more than 60 days. If you have been discharged from the hospital, the end of treatment visit will take place within 7 -14 days of the last day of study drug. You will need to return for the visit on an outpatient basis.

At this visit, you will have a physical exam, including measurement of vital signs (heart rate, temperature, and blood pressure). Blood samples (about 1 tablespoon) will be drawn for routine test and to check for infection. The blood sample may be drawn from the CVC, if the CVC is still in place. The CVC exit site will be examined. You will be asked about any symptoms or illnesses that you may have experienced. In addition, you will be asked to inform the study doctor and/or study staff of any medications or therapies that you are taking.

You will have a follow-up exam between 32 (+/- 7) days after your last dose of study drug. You will have a physical exam, including measurement of vital signs (heart rate, temperature, and blood pressure). Blood (about one tablespoon) will be drawn for routine tests and to check for infection. The blood samples may be drawn from the CVC, if the CVC is still in place. The CVC exit site may be examined. You will be asked about any symptoms or illnesses that you may have experienced. In addition, you will be asked to inform the study doctor and/or study staff of any medications or therapies that you are taking. Participation on this study will end once you complete the follow-up visit.

This is an investigational study. Daptomycin is approved by the FDA for the treatment of skin and soft tissue infection. However, for the use described in this study and at this dose level, Daptomycin is authorized by the FDA for use in research only. About 50 patients will take part in this study. All will be enrolled at the University of Texas (UT) MD Anderson Cancer Center (MDACC).

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating females with an age of greater than or equal to 18 years.
2. The suspected culprit on exchangeable central venous catheter (CVC) is tunnel ( including implanted ports) or non-tunneled catheter, antibiotic or non-antibiotic coated catheter inserted in the subclavian, jugular or femoral vein.
3. Patients must have at least two signs of sepsis from the list below, in any combination, within 48 hours prior to Daptomycin therapy and no other source for the bacteremia other than CVC: (a) Core temperature =/>38.0 degrees C or =/<36.0 degrees C, measured orally, rectally, tympanically or via a central catheter. If axillary add 0.5 degrees C to the measured temperature; (b) Pulse rate =/> 100 beats/min.; (c) Respiratory rate =/> 20/min; (d) white blood count (WBC) count =/>12,000/mm^3 or =/<4,000/mm^3 differential count showing >10% band forms; (e) Systolic blood pressure=/ <90 mm Hg
4. Patients with suspected or definite diagnosis of uncomplicated CVC-related gram-positive bacteremia that includes at least one positive blood culture for S aureus. (If the positive blood culture is drawn through the CVC, then at least >15 colonies/ml will be required or the differential time of positive (DTP) of CVC at least 2 hours earlier than the peripheral culture)
5. Signed informed consent
6. No apparent source for the clinical manifestation of bacteremia other than the catheter

Exclusion Criteria:

1. Creatinine clearance <30 mL/min at the time gram positive bacteremia was diagnosed unless the patient is on dialysis
2. Bilirubin >4 times the upper limit of normal at the time gram positive bacteremia was diagnosed
3. Treatment with an antibiotic effective against Gram-positive bacterial infections for more than 48 hours within 72 hours of study medication initiation, unless treatment failed.
4. Documented S. aureus bacteremia within last 3 months due to source other than CVC.
5. Patients who have participated in another investigational anti-infective study within 30 days
6. History of hypersensitivity to lipopeptides
7. Presence of additional source of infection with same organism cultured from blood, eg. endocarditis (as evidenced by vegetations on an echocardiogram), septic thrombosis
8. Conditions with markedly decreased albumin in plasma (<1.5 g/dl), e.g., cirrhosis, nephritic syndrome, end-stage renal disease
9. Anticipated prolonged therapy >4 weeks
10. Prosthetic endovascular material
11. Oliguria defined as urine output of <20 cc/hour averaged over 24 hours.
12. Possible complicated CRBSI with persistent bacteremia for more than 48 hours on active antimicrobial therapy (such as osteomyelitis, endocarditis, and septic thrombosis.)
13. Evidence of catheter site purulence as evidenced by purulent discharge.
14. Patients with diagnosis of pneumonia that is related to S. aureus organism
15. Patients taking concomitant "statins" (HMG-CoA reductase inhibitors)
16. creatine phosphokinase (CPK) >10 times max-normal in asymptomatic patients and CPK >5 max-normal in symptomatic patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Clinical Response Rate | 7 weeks
  Clinical response of Daptomycin administered for treatment of catheter-related bloodstream infections due to Staphylococcus Aureus bacteria, evaluated within 7 weeks of initiating Daptomycin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Issam Raad, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org